CLINICAL TRIAL: NCT06130007
Title: 替雷利珠单抗联合含铂双药新辅助治疗用于提高可切除局部晚期口腔鳞癌下颌骨保留的前瞻性、单臂Ⅱ期临床试验
Brief Title: A Prospective, Single-arm Phase II Clinical Trial of Tislelizumab Combined With Platinum Doublet Neoadjuvant Therapy to Improve Mandibular Preservation in Resectable Locally Advanced Oral Squamous Cell Carcinoma.
Acronym: B2023-153
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuekui Liu (Other)
Responsible Party: Sponsor-Investigator, Xuekui Liu, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-153
Record Dates: First submitted 2023-10-17; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Clinical Protocols; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment with Trastuzumab in Combination with Platinum-Based Doublet (Experimental): A first-line chemotherapy regimen for oral squamous cell carcinoma involves combining paclitaxel with platinum agents. PD-1 antibodies have shown promise in cases where the cancer has recurred, metastasized, or didn't respond to platinum-based treatments. Research is ongoing on using immune induction therapy with surgery or chemoradiotherapy for locally advanced, resectable oral squamous cell carcinoma. Trastuzumab, in combination with standard chemotherapy, is being explored as an induction treatment for patients needing mandibulectomy due to tumor proximity to the mandible. This study is a prospective, single-arm, single-center Phase II explora.
  Interventions: Drug: Three-Week Treatment Regimen with Trastuzumab in Combination with Docetaxel and Platinum Triple Therapy

INTERVENTIONS:
Drug: Three-Week Treatment Regimen with Trastuzumab in Combination with Docetaxel and Platinum Triple Therapy — Three-Week Treatment Regimen with Trastuzumab in Combination with Docetaxel and Platinum Triple Therapy

SUMMARY:
Given the feasibility of induction chemotherapy in oral cancer and the encouraging remission rates achieved, we explore the clinical application prospects of using tislelizumab in combination with traditional standard chemotherapy as induction treatment in oral cancer patients who have no radiological evidence of mandibular erosion but require mandibulectomy due to the tumor's proximity to the mandible, aiming to shrink tumor size and increase the rate of mandible preservation. Therefore, we propose to conduct a prospective, single-arm, single-center phase II exploratory clinical trial: we plan to select patients with locally advanced resectable primary oral squamous cell carcinoma T3-4N0-3M0 (stages III-IVb, excluding T1-2) after multidisciplinary consultation and assessment by imaging and clinical evaluation. We aim to explore the feasibility of a three-week treatment regimen combining tislelizumab with polyaletin paclitaxel and a platinum-based triplet, preliminarily assess its clinical efficacy, adverse reactions, and postoperative mandible preservation rate, to provide the best comprehensive treatment plan for the preservation rate of the mandible in oral squamous cell carcinoma.

DETAILED DESCRIPTION:
In this study, eligible subject will be enrolled into study arm to accept study treatment mandibular Preservation Rate will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Patients must have a confirmed diagnosis of untreated primary oral squamous cell carcinoma, originating from the buccal mucosa, gums, tongue, or floor of the mouth, with clinical imaging confirming no mandibular invasion. Even in the absence of mandibular invasion, patients must still require mandibular segment resection.

Clinical staging should be T3-4N0-3M0 (Stage III-IVb, excluding T1-2) according to the AJCC 8th edition staging.

Patients must be aged between 18 and 70 years. Performance Status (PS) score should be 0-1. Evaluation by a head and neck oncologist should confirm eligibility for surgical resection.

Patients should have at least one evaluable lesion according to RECIST V1.1 criteria.

Adequate organ function is defined as follows:

Hematology: White blood cells ≥ 4000/μL, neutrophils ≥ 2,000/μL, hemoglobin ≥ 90 g/dL, platelets ≥ 100,000/μL.

Liver function: Bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert's disease and serum bilirubin levels ≤ 3 times ULN may be eligible), AST and ALT ≤ 3 times ULN, and alkaline phosphatase ≤ 3 times ULN, with albumin ≥ 3 g/dL.

Renal function: Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula.

Coagulation parameters (APTT and INR) should be ≤ 1.5 × ULN (patients on stable anticoagulation therapy such as low molecular weight heparin or warfarin within the expected therapeutic range may be screened).

Thyroid-stimulating hormone (TSH) should be ≤ ULN. If abnormal, T3 and T4 levels should be assessed, and patients with normal T3 and T4 levels may be eligible.

Patients must have provided informed consent and must be willing and able to adhere to the study plan, visit schedule, treatment plan, laboratory tests, and other study procedures.

Reproductive-age females must agree to use contraceptive measures (e.g., intrauterine device, birth control pills, or condoms) during the treatment period and for three months after treatment completion. A negative serum or urine pregnancy test within 7 days before study entry is required, and patients must not be breastfeeding. Male patients must also agree to use contraceptive measures during the study and for three months after study completion.

Exclusion Criteria:

* Exclusion Criteria:

History of severe hypersensitivity reactions to other monoclonal antibodies or PD-1 monoclonal antibodies or any of their components.

Known or suspected autoimmune diseases, including dementia and epileptic seizures.

Presence of measurable residual disease or new tumor/metastasis according to RECIST1.1 criteria, or patients deemed inoperable following evaluation by a head and neck specialist.

Abnormal coagulation function: (PT > 16s, APTT > 53s, TT > 21s, Fib < 1.5g/L), a tendency to bleed, or current treatment with thrombolytic or anticoagulant agents.

Severe cardiac or pulmonary dysfunction, with heart or lung function rated below Grade 3 (inclusive).

Abnormal laboratory values within 7 days before enrollment.

History of any of the following treatments:

1. Prior use of anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4 antibodies (or any other antibodies targeting T cell co-stimulatory or checkpoint pathways).
2. Receipt of any investigational drug within 4 weeks before the first dose of the study drug.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or a follow-up study for a new clinical trial.
4. Pre-existing conditions requiring long-term use of immunosuppressive drugs or the use of corticosteroids at doses with immunosuppressive effects, either systemically or locally.
5. Vaccination with anti-tumor vaccines or receipt of live vaccines within 4 weeks before the first dose of the study drug.
6. Major surgery or severe trauma within 4 weeks before the first dose of the study drug.

Experienced severe infections (CTC AE Grade > 2) within 4 weeks before the first use of the study drug, such as severe pneumonia, septicemia, or complications of infection requiring hospitalization; baseline chest imaging indicating active lung inflammation; presence of symptoms and signs of infection within 2 weeks before the first use of the study drug or the need for oral or intravenous antibiotics (excluding prophylactic antibiotic use).

HIV-positive individuals, those testing positive for HBsAg with concurrent detection of positive HBV DNA copy numbers (quantitative test ≥ 1000 cps/ml); positive screening for chronic hepatitis C (HCV antibody-positive).

History of other malignant tumors in the past 5 years, except for cured basal cell carcinoma, in situ cervical carcinoma, and papillary thyroid carcinoma.

Positive pregnancy test in women of childbearing age and breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Mandibular Preservation Rate; | 12 weeks
  Mandibular Preservation Rate

SECONDARY OUTCOMES:
ORR | 12 weeks
  Objective Response Rate
CR | 12 weeks
  Complete Response
PR | 12 weeks
  Partial Response
SD | 12 weeks
  Stable Disease
PD | 12 weeks
  Disease Progression
MPR | 12 weeks
  major pathological response
pCR | 12 weeks
  complete pathological response rate
PFS | 3 years
  progression-free survival
DFS | 3 years
  disease-free survival
OS | 3 years
  overall survival
AE | 90 days after the first dose of study treatment
  Percentage of adverse events that are possibly, probably related to study treatment per Criteria for Adverse Events version 5(CTCAE v5.0)

IPD SHARING:
Plan to Share IPD: No